CLINICAL TRIAL: NCT06820437
Title: Comparison of the Effectiveness of High-Fidelity Simulation and Low-Fidelity Simulation in the Management of Active External Bleeding Control by Caregivers of Elderly Individuals
Brief Title: Comparison of the Effectiveness of High Fidelity Simulation and Low Fidelity Simulation in Active External Bleeding Control Management of Caregivers of Elderly Individuals
Status: Not yet recruiting | Type: Observational
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Songül Demir, Doctorate Student- Lecturer, Mustafa Kemal University
Other Study IDs: 2023/16
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Simulation Training; High Fidelity Simulation Training; First Aid; Informal Caregivers; Elderly; Bleeding
Keywords: Elderly caregivers; external bleeding; elderly; first aid training; simulation; visually enhanced mental simulation; high fidelity simulation
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group 1:: VEMS (low-fidelity simulation)
  Interventions: Other: Low-fidelity (Visually Enhanced Mental Simulation-VEMS) simulation training
- Intervention group 2: High-fidelity (simulated patient/standard patient) simulation
  Interventions: Other: High-fidelity (simulated patient/standard patient) simulation training

INTERVENTIONS:
Other: Low-fidelity (Visually Enhanced Mental Simulation-VEMS) simulation training — Intervention group 1: Low-fidelity (Visually Enhanced Mental Simulation-VEMS) simulation training will be conducted on active external bleeding control management skills of caregivers of elderly individuals. In this intervention poster and cards will be used.
  Groups: Intervention group 1:
Other: High-fidelity (simulated patient/standard patient) simulation training — Intervention group 2: High-fidelity (simulated patient/standard patient) simulation training will be conducted for caregivers of elderly individuals in active external bleeding control management skills. Standardized patient who will act as elderly will be used in this intervention.
  Groups: Intervention group 2

SUMMARY:
The elderly population is increasing worldwide. Due to the increase in the elderly population, emergencies related to ageing are also encountered more frequently. One of these emergencies is trauma in the elderly. Traumas are frequently seen in elderly individuals due to physiological deficiencies related to aging as well as environmental factors. External bleeding caused by trauma is also encountered. If first aid to stop active external bleeding is not administered in a timely and correct manner, death due to bleeding can occur. Nowadays, elderly individuals live either with their families, alone, or in institutions. In the event of external bleeding, either the individual themselves, caregiving family members, or staff at the institution should be able to perform first aid to stop the bleeding.

Elderly individuals may not be able to perform first aid due to cognitive and neurological deficiencies. The ability of caregivers to provide first aid can be life-saving. If caregivers of elderly individuals are trained in first aid for external bleeding, they can quickly and correctly administer first aid to stop the bleeding. First aid training often consists of didactic education and demonstrations. A training strategy that ensures knowledge retention and skill acquisition is simulation training. This study aims to evaluate and compare the effectiveness of high-fidelity simulation and low-fidelity (Visually Enhanced Mental Simulation - VEMS) simulation in the skills of caregivers for elderly individuals in managing active external bleeding control.

The population of the study will consist of non-health professional caregivers of elderly individuals living in Antakya district of Hatay province. The sample size, calculated using the G Power program, has been determined to include 30 caregivers of elderly individuals. The study consists of four main work packages. In the first stage, the simulation environment will be prepared, and in the second stage, a preliminary application of the project will be conducted. In the third stage, the implementation of the research and the completion of checklists will be ensured. For this, volunteer caregivers of elderly individuals will be identified. After theoretical training is given to the participants, they will be assigned to intervention group 1 (VEMS) and intervention group 2 (high-fidelity simulation) using simple randomization. Following a pre-assessment with low-fidelity simulation, participants will undergo simulation training according to their intervention groups. Subsequently, a final assessment will be conducted using the same lowfidelity simulation. In the final stage, data analysis and interpretation of the findings will be carried out. The collected data will be analyzed statistically, and the significance level will be accepted as p<0.05. With this study, insight will be provided into the effectiveness of VEMS and high-fidelity simulation in first aid training for active external bleeding for caregivers of elderly individuals. On the other hand, it is planned that the project results will be published in at least one article in journals indexed in the SSCI Expanded.

ELIGIBILITY:
Inclusion Criteria:

* Not having received the theoretical first assessment and first aid training in external bleeding
* No cognitive and communication problems that can actively participate in the study
* Not being a health professional
* Not being a paid caregiver

Exclusion Criteria:

* The participant declares that he/she wants to leave at any stage of the study
* Not participating in any of the simulation phases
* Not participating in the implementation of the data collection tools to be applied

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of the study will consist of non-health professional caregivers of elderly individuals living in Antakya district of Hatay province. The sample size was determined by calculating in the G Power program. With 95% confidence (1-α), 95% test power (1-β), d=1.387 effect size and two-way independent samples t-test, the number of samples to be taken in each group was determined as 15 (Scalese et al., 2022). After the theoretical training, participants will be randomly assigned to groups by lottery method. With the support of neighborhood mukhtars, individuals who care for elderly individuals will be contacted and informed about the study, and volunteer caregivers who are not health professionals will be included in the study by signing informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Active external bleeding control management skills of caregivers of elderly individuals assesed by "Active External Bleeding Management Asssesment Form" | 1st - 4 th months
  Active External Bleeding Management Asssesment Form was developed by the researchers. It includes 13 items which evaluate first aid inteventions for external bleeding. Expert opininons were taken for content validity of the form.

SECONDARY OUTCOMES:
Obtaining the opinions of caregivers of elderly individuals on the interventions by using Simulation Assesment Form | 1st-4th months
  The opinions of the caregivers of elderly individuals about the interventions, which are high fidelity simulation and low fidelity simulation in active external bleeding control management skills, will be obtained through questionnaires developed by the researchers in the light of the literature by taking expert opinion. The form includes likert type 12 items.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Hatay Mustafa Kemal University, Hatay, Antakya
  - Hatay Mustafa Kemal University, Antakya, Hatay

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abou-Raya S, ElMeguid LA. Road traffic accidents and the elderly. Geriatr Gerontol Int. 2009 Sep;9(3):290-7. doi: 10.1111/j.1447-0594.2009.00535.x. PMID 19702940
- [Background] Abatzis VT, Littlewood KE. Debriefing in Simulation and Beyond. Int Anesthesiol Clin. 2015 Fall;53(4):151-62. doi: 10.1097/AIA.0000000000000070. PMID 26397791